CLINICAL TRIAL: NCT03410264
Title: One-session Treatment for Spider Fears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1609
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-02

CONDITIONS: Spider Phobia
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with three treatment conditions.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CR-EXP (Experimental): Cognitive restructuring before exposure with response prevention (45 minute intervention).
  Interventions: Behavioral: CR-EXP
- EXP-CR (Experimental): Exposure with response prevention before cognitive restructuring (45 minute intervention).
  Interventions: Behavioral: EXP-CR
- Stress Management (Active Comparator): Stress management skills.
  Interventions: Behavioral: Stress Management

INTERVENTIONS:
Behavioral: CR-EXP — See arm/group descriptions
  Arms: CR-EXP
Behavioral: EXP-CR — See arm/group descriptions
  Arms: EXP-CR
Behavioral: Stress Management — See arm/group descriptions
  Arms: Stress Management

SUMMARY:
Despite the efficacy of exposure and response prevention (ERP) for anxiety and phobias, recent theoretical research on fear extinction via inhibitory learning suggests that cognitive restructuring (CR)--the explicit challenging of maladaptive beliefs (e.g,. overestimation of threat)--may actually attenuate exposure outcomes during an exposure trial. That is, by verbally disputing certain beliefs (e.g., "the spider will jump on me and attack me and I will faint from the anxiety") before an exposure task (e.g., gradually approaching a non-venomous spider), anxious individuals may experience less "surprise" from the non-occurrence of feared outcomes, and consequently experience less inhibitory learning (e.g., learning that spiders are not inherently dangerous). Thus, the investigators aim to empirically test the conventional (yet recently challenged) assumption that cognitive restructuring is a necessary component for psychosocial interventions for phobias.

90 participants recruited from the Psychology Department Participant Pool and the community will participate in this study. All participants will meet DSM-5 criteria for spider phobia. Following consent, participants will complete a pre-test assessment of various aspects of spider phobia. Participants will then receive education about the nature of anxiety/spider phobia and be randomly assigned to one of three 45-min intervention conditions: (a) CR before EXP, (b) EXP before CR, and (c) stress management (a control condition that involves neither CR nor EXP). Following the intervention, participants will complete a 10-minute post-test assessment and be scheduled to return for a follow-up assessment a month later.

DETAILED DESCRIPTION:
Recent conceptualizations of the mechanisms by which exposure therapy (EXP; i.e., confronting one's fear in a systematic and therapeutic way) works in the treatment of phobias focus on the importance of extinction learning). This "inhibitory learning model" proposes that EXP helps the phobic individual learn that phobic stimuli are not dangerous; yet older danger-related learning is not "erased", and so must be inhibited by the new "safety learning." Research indicates that incorporating surprise into EXP (e.g., the patient is surprised that the spider didn't bite) maximizes this type of inhibitory learning and would correspond to better outcomes for phobias then when there is no surprise at the outcome of EXP.

Traditionally, EXP is used with the addition of cognitive restructuring (CR), which involves discussing and disputing exaggerated beliefs that underlie one's fears (e.g., "spiders are very dangerous"). CR encourages phobic individuals to re-evaluate their expectations of danger when encountering phobic stimuli, and therefore might rob the individual of the opportunity to be surprised when actually facing their fear.

Despite the theoretical plausibility of the importance of surprise during EXP, this question has yet to be investigated empirically. The aim of the present study is to test the hypothesis that incorporating surprise into EXP (by postponing CR until after EXP) will enhance immediate and long-term outcome of EXP for spider phobia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must

  1. be 18 years or older,
  2. be fluent in English, and
  3. meet DSM-5 criteria for specific (spider) phobia to be considered eligible

Exclusion Criteria:

* Participants will be deemed ineligible if they do not meet the above inclusion criteria or

  1. are allergic to spiders or bee stings,
  2. are experiencing current psychosis, mania, or substance abuse, or
  3. successfully complete 10 of 13 possible BAT steps in the pretreatment appointment (to ensure that participants are indeed spider phobic at pretreatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Behavioral Approach Task (BAT) at 1-month follow-up | Baseline, 1-month follow-up
  The Behavioral Approach Task (BAT) includes 13 rank-ordered steps ranging from standing at the opposite end of a room containing a tarantula enclosed in a closed terrarium covered with a sheet to allowing the tarantula to crawl up one's bare arm. A participant must perform a BAT step for 10 consecutive seconds for the step to count as completed. BAT scores are recorded as the number of the highest step completed. Immediately after completing each step of the BAT (at the baseline and post-treatment assessments), participants are asked to verbally report their (a) anxiety and (b) disgust, using a scale of 0 (not at all) to 10 (maximum).
Change from baseline Spider Beliefs Questionnaire (SBQ) at 1-month follow-up | Baseline, 1-month follow-up
  The SBQ is a 78-item scale measuring one's concerns related to encounters with spiders. Items are rated on a 0-100 scale (0= I do not believe it at all (0%); 100= I absolutely believe it (100%)). Total scores range from 0-7800. Higher scores indicate more negative beliefs about spiders.
Change from baseline Spider Self-Efficacy Scale (SSES) at 1-month follow-up | Baseline, 1-month follow-up
  The Spider Self-Efficacy Scale (SSES) is a self-report measure of the strength of self-efficacy about performing behaviors related to spiders. The scale consists of 26 items describing approach behaviors towards spiders, on which respondents rate the strength of their self-efficacy about performing that behavior on an 11-point scale ranging from 0 (no confidence/highly uncertain) to 10 (total confidence/complete certainty). Total scores range from 0 to 260. Higher scores indicate higher self-efficacy.

SECONDARY OUTCOMES:
Change from baseline Distress Tolerance Scale (DTS) at 1-month follow-up | Baseline, 1-month follow-up
  The DTS is a 15-item self-report measure of one's ability to tolerate psychological distress. Items are rated on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree). Total scores range from 15 to 75. High scores on the DTS indicate that an individual can tolerate high levels of distress. Low scores reflect low DT (i.e., distress intolerance).
Change from baseline Distress Tolerance Scale (DTS) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The DTS is a 15-item self-report measure of one's ability to tolerate psychological distress. Items are rated on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree). Total scores range from 15 to 75. High scores on the DTS indicate that an individual can tolerate high levels of distress. Low scores reflect low DT (i.e., distress intolerance).
Change from baseline Anxiety Sensitivity Index-3 (ASI-3) at 1-month follow-up | Baseline, 1-month follow-up
  The ASI is a 16-item self-report measure of beliefs regarding the dangerousness of anxious arousal (e.g., "It scares me when my heart beats rapidly"). Participants rate their agreement with each statement on a 0 (very little) to 4 (very much) scale; higher scores indicate greater anxiety sensitivity. Total scores range from 0 to 64.
Change from baseline Anxiety Sensitivity Index-3 (ASI-3) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The ASI is a 16-item self-report measure of beliefs regarding the dangerousness of anxious arousal (e.g., "It scares me when my heart beats rapidly"). Participants rate their agreement with each statement on a 0 (very little) to 4 (very much) scale; higher scores indicate greater anxiety sensitivity. Total scores range from 0 to 64.
Change from baseline Depression Anxiety Stress Scales-21 (DASS-21) at 1-month follow-up | Baseline, 1-month follow-up
  The DASS-21 is a 21-item self-report measure of general psychological distress. Participants rate items on a four-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time). Total scores range from 0 to 63, and higher scores indicate more distress.
Change from baseline Depression Anxiety Stress Scales-21 (DASS-21) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The DASS-21 is a 21-item self-report measure of general psychological distress. Participants rate items on a four-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time). Total scores range from 0 to 63, and higher scores indicate more distress.
Change from baseline Disgust Scale-Revised (DS-R) at 1-month follow-up | Baseline, 1-month follow-up
  The DS-R is a 25-item measure of respondents' propensity to experience disgust across multiple domains. Participants rate the degree to which they might find a number of scenarios (e.g., ''you see maggots on a piece of meat in an outdoor garbage pail'') disgusting on a scale of 0 (strongly disagree) to 4 (strongly agree). Total scores range from 0 to 100, and higher scores indicate more disgust sensitivity.
Change from baseline Disgust Scale-Revised (DS-R) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The DS-R is a 25-item measure of respondents' propensity to experience disgust across multiple domains. Participants rate the degree to which they might find a number of scenarios (e.g., ''you see maggots on a piece of meat in an outdoor garbage pail'') disgusting on a scale of 0 (strongly disagree) to 4 (strongly agree). Total scores range from 0 to 100, and higher scores indicate more disgust sensitivity.
Change from baseline Anxiety Control Questionnaire (ACQ) at 1-month follow-up | Baseline, 1-month follow-up
  The Anxiety Control Questionnaire (ACQ) comprises 30 items and assesses the perception of control over emotional reactions (e.g., "My emotions seem to have a life of their own") and external threats (e.g., "I am usually able to avoid threat quite easily"). This self-report instrument attributes lower scores to individuals with lower perceptions of control and provides. Participants respond on a 0-5 scale, and total scores range from 0 to 150.
Change from baseline Anxiety Control Questionnaire (ACQ) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The Anxiety Control Questionnaire (ACQ) comprises 30 items and assesses the perception of control over emotional reactions (e.g., "My emotions seem to have a life of their own") and external threats (e.g., "I am usually able to avoid threat quite easily"). This self-report instrument attributes lower scores to individuals with lower perceptions of control and provides. Participants respond on a 0-5 scale, and total scores range from 0 to 150.
Change from baseline Acceptance and Action Questionnaire-II (AAQ-II) at 1-month follow-up | Baseline, 1-month follow-up
  The Acceptance and Action Questionnaire-II (AAQ-II) is a 10-item revision of the original 9-item AAQ. Each item is rated from 1 (never true) to 7 (always true) and total scores range from 10 to 70. The scale assesses experiential avoidance, also known as ''psychological flexibility,'' which is a core construct of the acceptance and commitment therapy model of psychopathology. Higher scores on the AAQ-II indicate greater psychological flexibility (less pathology).
Change from baseline Acceptance and Action Questionnaire-II (AAQ-II) at 0-5 hours post-treatment | Baseline, 0-5 hours post-treatment
  The Acceptance and Action Questionnaire-II (AAQ-II) is a 10-item revision of the original 9-item AAQ. Each item is rated from 1 (never true) to 7 (always true) and total scores range from 10 to 70. The scale assesses experiential avoidance, also known as ''psychological flexibility,'' which is a core construct of the acceptance and commitment therapy model of psychopathology. Higher scores on the AAQ-II indicate greater psychological flexibility (less pathology).

CONTACTS AND LOCATIONS:
Overall Officials: Jon Abramowitz, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States